CLINICAL TRIAL: NCT00345709
Title: The Elizabeth Registry for Low Grade Ovarian Cancer
Brief Title: Elizabeth Registry for Low Grade Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0359
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Elizabeth Registry; Questionnaire; Registry; Survey
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- National Research Registry Enrollment: Patient, living or deceased, with a pathologically-confirmed diagnosis of Ovarian Cancer.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 65 page questionnaire that contains questions about your ovarian cancer diagnosis, gynecologic history, family history, general medical history, and health risk factors.
  Other Names: Survey

SUMMARY:
Long-Term Objectives:

* To establish an ongoing national research registry of epidemiologic, clinical and pathologic data on low grade and low malignant potential (LMP) ovarian cancer patients in UTMDACC's Department of Gynecologic Oncology for research purposes.
* To create a bank of low grade and LMP ovarian cancer tumor blocks for study of the molecular and histopathologic differences among low grade ovarian cancer, ovarian LMP tumors and high grade ovarian cancer.
* To specify the epidemiologic and clinical profile of low grade and LMP ovarian cancer patients.
* To identify potential precursors of low grade and LMP ovarian cancer.
* To assess treatment patterns to guide management of these diseases.
* To collect quality of life and health outcomes data on these patients.
* To achieve a fundamental understanding of low grade and LMP ovarian cancer that will inform prevention and screening efforts, motivate development of improved treatments and eventually result in a cure.

The short-term objectives are:

* To detail procedures for potential registrant identification and recruitment.
* To create a demographic and health history questionnaire for potential registrants.
* To begin aggregating low grade and low malignant potential ovarian tumor blocks.
* To specify a timeline for the development of all other aspects of the Registry.

DETAILED DESCRIPTION:
The Registry will be an ongoing research registry that will include patients who have been diagnosed with low grade ovarian, primary peritoneal or fallopian tube or low malignant potential (LMP) ovarian, primary peritoneal or fallopian tube cancer.

In order to enroll in the Registry, you will be asked to complete a 65 page questionnaire that contains questions about your ovarian cancer diagnosis, gynecologic history, family history, general medical history, and health risk factors. This questionnaire will take about 1 hour to complete.

In addition, researchers will look at your medical record and pathology samples stored at M. D. Anderson to get information about your surgeries, treatments, disease course, and tumor grade. If your original surgery was not performed at M. D. Anderson, you may be asked to provide tumor specimens from that surgery before enrolling in the Registry.

You will be contacted annually by the Registry Coordinator to update your demographic and health information.

This is an investigational study. The Registry will eventually enroll both M. D. Anderson and non-M. D. Anderson patients. The number of registrants is unlimited because the Registry will be ongoing. This study is partially funded by a research grant from the Elizabeth Fund for the Study of Low Grade Ovarian Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. UTMDACC patient, living or deceased, with a pathologically-confirmed diagnosis of either low grade ovarian carcinoma or LMP ovarian carcinoma.
2. Able to speak and read English (for patients who are living).
3. Residence in the United States, both at time of original diagnosis and at time of accession to the Registry.

Exclusion Criteria:

1. UTMDACC patients, living or deceased, whose diagnosis of either low grade ovarian carcinoma or LMP ovarian carcinoma has not been confirmed pathologically.
2. Any type of ovarian cancer other than low grade or LMP ovarian carcinoma.
3. Unable to speak and read English (for patients who are living).
4. Residence outside the United States, either at time of original diagnosis or at time of accession to the Registry.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: M.D. Anderson Cancer Center Patient, living or deceased, with a pathologically-confirmed diagnosis of either low grade ovarian carcinoma or LMP ovarian carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Establish an ongoing national research registry of epidemiologic, clinical and pathologic data on low grade and low malignant potential (LMP) ovarian cancer patients in UTMDACC's Department of Gynecologic Oncology for research purposes. | 30 Years

SECONDARY OUTCOMES:
Create a bank of low grade and LMP ovarian cancer tumor blocks for study of the molecular and histopathologic differences among low grade ovarian cancer, ovarian LMP tumors and high grade ovarian cancer. | 30 Years
Specify the epidemiologic and clinical profile of low grade and LMP ovarian cancer patients. | 30 Years
Identify potential precursors of low grade and LMP ovarian cancer. | 30 Years
Assess treatment patterns to guide management of these diseases. | 30 Years
Collect quality of life and health outcomes data on these patients. | 30 Years

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org